CLINICAL TRIAL: NCT01686776
Title: A Prospective Validation Study in Healthy Volunteers, Patients With Acute Inflammation and Patients Scheduled for Major Abdominal Surgery
Brief Title: A Prospective Validation Study of Albumin Kinetics With Tracer 123 I-HSA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ake Norberg (Other)
Responsible Party: Sponsor-Investigator, Ake Norberg, M.D, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3.00 # amended version 1.1; 2012-002638-35 (EudraCT Number)
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Healthy; SIRS
Keywords: Plasma albumine; Plasma volume; Transcapillary escape rate; Inflammation; Circulation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: 3 parallell Groups were measured regarding plasma volume and transcapillary escape rate of albumin where commercial 125I-iodinated human serum albumin was compared to hospital manufactured 123I- iodinated human serum albumin
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 123 I-HSA + 125 I-HSA (Active Comparator): Healthy Volunteers, N=16
  Interventions: Other: 123 I-HSA + 125 I HSA
- 123 I- HSA + 125 I-HSA (Experimental): Patients, planned for elective Major Abdominal Surgery, N=16
  Interventions: Other: 123 I-HSA + 125 I HSA
- 123-I-HSA+125 I-HSA (Experimental): Patients, with a acute pancreatitis or cholecystitis, N=16
  Interventions: Other: 123 I-HSA + 125 I HSA

INTERVENTIONS:
Other: 123 I-HSA + 125 I HSA — Compare and validate the method of measuring albumine turnover rate

SUMMARY:
This is a prospective, validation study of a extempore made tracer compared with a commercial. Studies with tracer have no medical effects but are used for studying human physiology, in this case pharmacokinetic variables of endogenous albumin distribution and turnover at different levels of inflammation.

1. Primary Objective:

   - Do the extempore made tracer 123-iodine labeled albumin an commercially manufactured SERALB-125 give identical values of calculated blood plasma volume and capillary leakage measured as transcapillary escape rate of albumin?
2. Secondary Objective:

   * How do three different measures of albumin turnover correlate in volunteers?
   * How do the pharmacokinetic parameters of endogenous albumin vary between the three study groups?

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (treatment arm I)
* on contraceptive agent and/or contraceptive device
* visual peripheral veins
* signed informed consent
* planned for elective larger interabdominal surgery (treatment arm II)
* patients with a acute pancreatitis or cholecystitis (treatment arm III)

Exclusion Criteria:

* pregnant women and/or lactating
* allergy towards excipients in 123 I HSA or 125 I HSA
* participates in another study involving radiation or stabile isotopes within a period of 60 days to study start
* it is the opinion of the principle investigator that the patient/subject should not participate for his/hers own good

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Transcapillary Escape Rate (TER)of Albumin | 42 days
  Is the measured value for 123-I-HSA and 125I-HSA identical/equal regarded TER and plasma volume (PV)?

SECONDARY OUTCOMES:
Fractional catabolic rate (FCR) | 42 days
  Non compartmental analysis (NCA) and AUC (time-conc) will be determine the pharmacokinetics like clearance, distribution volume and absolute catabolic rate

OTHER OUTCOMES:
plasma albumin turnover rate | 42 days
  How well does the variables FSR, FCR1, FCR30 correlate? How does the pharmacokinetic parameters differ/varies between the three groups?

CONTACTS AND LOCATIONS:
Overall Officials: Olav Rooyackers, PhDProfessor, Study Chair — Karolinska University Hopsital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Result] Komaromi A, Estenberg U, Hammarqvist F, Rooyackers O, Wernerman J, Norberg A. Simultaneous assessment of the synthesis rate and transcapillary escape rate of albumin in inflammation and surgery. Crit Care. 2016 Nov 15;20(1):370. doi: 10.1186/s13054-016-1536-6. PMID 27846908